CLINICAL TRIAL: NCT01556360
Title: Bone Status on Patients With Genetic Hemochromatosis : a 3 Years Descriptive and Evolutionary Study.
Brief Title: Bone Status on Patients With Genetic Hemochromatosis: a 3 Years Descriptive and Evolutionary Study
Acronym: FEROS
Status: Completed | Type: Observational
Sponsor: Rennes University Hospital (Other)
Collaborators: Ministry of Health, France (Other Government)
Responsible Party: Sponsor
Other Study IDs: 2008-A000386-47
Record Dates: First submitted 2012-03-01; First posted 2012-03-16 (Estimated); Last update posted 2015-05-27 (Estimated); Status verified 2015-05

CONDITIONS: Genetic Hemochromatosis
Keywords: genetic hemochromatosis; Iron overload; C282 homozygosity
MeSH Terms: conditions — Hemochromatosis; Iron Overload

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — * serum
  * urine
  * DNA
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to describe bone status on patients with genetic hemochromatosis, at diagnostic time and his evolution under treatment.

DETAILED DESCRIPTION:
Bone diseases have been recognized recently as complications of genetic hemochromatosis. Further studies are needed to describe the role of iron in bone injuries. The purpose of this study is to describe bone status on patients with genetical hemochromatosis, at diagnostic time and his evolution under treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patients between 18 and 80 years
* C282 homozygosity

Exclusion Criteria:

* corticosteroids during the last 3 months
* following treatments during the last 6 months : anabolic steroids, growth hormone, hormone therapy for menopause, tibolone, raloxifene.
* following treatments during inclusion or in the last 6 month : teriparatide, parathormone, fluor, strontium ranelate, biphosphonate.
* cancer or evolutionary hemopathy (including monoclonal gammopathy)
* pregnancy at inclusion time
* treated osteoporosis
* patient in wich follow up seems hard
* inclusion in another study incompatible with this one

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient with genetic hemochromatosis diagnosed in western France hospitals
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2008-07; Primary Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Bone mineral density | Change from baseline in bone mineral density at three years
  Vertebral and hips Dual energy X-ray Absorptiometry (DXA)

SECONDARY OUTCOMES:
Predictive value of iron overload on Bone Mineral Density | 1 day
Number of vertebral fractures | 3 years
Number of peripheral fractures | 3 years
Number and location of joint lesions detected by the examination (pain and swelling) | 3 years
Determination of genetic polymorphism of BMP 2 and 4 | Baseline

CONTACTS AND LOCATIONS:
Overall Officials: Guggenbuhl Pascal, MD, Principal Investigator — Rennes University Hospital
Locations (6):
- France (6):
  - Angers University Hospital, Angers
  - Brest University Hospital, Brest
  - Nantes University Hospital, Nantes
  - Orleans Regional Hospital, Orléans
  - Poitiers University Hospital, Poitiers
  - Rennes University Hospital, Rennes